CLINICAL TRIAL: NCT06756425
Title: Effect of Aerobic Exercise Program on Blood Glucose Level and Quality of Life in Pre-diabetic Overweight/Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marina Nabil Samaan Meseha, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005129
Record Dates: First submitted 2024-12-14; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Prediabetes
Keywords: obesity; prediabetes; aerobic exercises; quality of life; blood glucose level; HbA1C; adolescents
MeSH Terms: conditions — Obesity; Prediabetic State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group, overweight and obese adolescents with prediabetes (Active Comparator)
  Interventions: Behavioral: aerobic exercise program; Behavioral: nutritional health awareness sessions
- control group, overweight and obese adolescents with prediabetes (Active Comparator)
  Interventions: Behavioral: nutritional health awareness sessions

INTERVENTIONS:
Behavioral: aerobic exercise program — aerobic exercise program for 3 months with nutritional health awearness sessions
  Arms: study group, overweight and obese adolescents with prediabetes
Behavioral: nutritional health awareness sessions — lifestyle changes and nutritional awareness sessions for 3 months twice a week for participants and their parents

SUMMARY:
PURPOSE:

The study aims to:

Investigate the effect of the designed aerobic exercise program on the blood glucose level (fasting blood glucose and HbA1C) in overweight/ obese pre-diabetic adolescents.

2) Investigate the effect of the designed aerobic exercise program on the BMI, aerobic capacity, and waist circumference of the participant before and after the designed aerobic exercise program.

3) Investigate the effect of the designed aerobic exercise program on the quality of life in overweight/ obese pre-diabetic adolescents.

4) Compare the effect of the diet program only and the diet with a designed aerobic exercise program on the blood glucose level (FBG, HbA1C) and the quality of life of the participants.

BACKGROUND:

Obesity is defined as a common chronic disorder of excessive body fat. It has become a global epidemic that is present not only in the industrialized world but also in many developing and even underdeveloped countries (Hans, 2017).

Overweight children and adolescents often suffer from symptoms of depression and anxiety, poor self-esteem, and social stigma. These psychological aspects complicate global care and affect the quality of life (QOL). The overall QOL score was lower in the overweight and obese groups compared with the normal-weight groups in all the clinical population studies. The published results also indicate that impairment in QOL worsens with a degree of obesity (Marie et al., 2014).

HYPOTHESES:

There will be no significant difference effect between the diet program only and diet program with a designed aerobic exercise program on blood glucose levels and QOL in overweight/ obese prediabetic adolescents.

RESEARCH QUESTION:

Does the designed aerobic exercise influence the blood glucose level and the quality of life in pre-diabetic overweight/obese adolescents?

ELIGIBILITY:
Inclusive criteria:

The participants will be selected according to the following criteria:

1. Their ages range from 12 to 18 years old.
2. They will be overweight and obese according to BMI charts of CDC:

   * Overweight is 85 percentiles to less than the 95 percentile,
   * Obesity is 95 percentile or greater) (CDC, 2022).
3. They will be prediabetic according to CDC, USPSTF (2022):

   * HbA1c level of will be 5.7% to 6.4%,
   * A fasting plasma glucose level will be 100 to 125 mg/dL.
4. Their waist circumference percentiles will be in the area outside of the normal WC curve according to WHO, normal children and adolescents are in the area under the curve (AUC): 0.69 for boys; 0.63 for girls for normal adolescents) (Bo xi et al., 2020)
5. They will be able to follow instructions during evaluation and treatment.

Exclusive criteria:

Any adolescent with the following criteria will be directly excluded from the evaluation for the consistency of the sample and statistically obtained results:

1. Cardiovascular diseases,
2. Diabetes Mellitus,
3. Morbid obesity more than 120% of the 95 percentile or greater or 35 kg/m or greater.
4. Hearing or visual impairments.
5. Any orthopedic deformities in upper limb or lower limb.
6. Uncontrolled seizures.
7. Receiving any special medications.
8. Participated regularly in sportive activities.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
changed HbA1c | 3 months
changed BMI | 3 months
changed Quality of life questionnaire results | 3 months

SECONDARY OUTCOMES:
changed waist circumference | 3 months
changed fasting blood glucose level | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided